CLINICAL TRIAL: NCT07118865
Title: Assessing the Impact of Internet-Guided Pilates Training on People With Hypermobility
Brief Title: Online Pilates Exercise for People With Hypermobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarkson University (Other)
Responsible Party: Principal Investigator, Leslie Russek, Professor Emeritus of Physical Therapy, Clarkson University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-48.3
Record Dates: First submitted 2025-07-30; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome; Hypermobile Spectrum Disorder
Keywords: hypermobile Ehlers-Danlos Syndrome, Pilates, Exercise
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was a pragmatic clinical trial with an intervention group and a wait-list control group. The groups were assigned sequentially and not randomly: the first group of about 300 subjects was allowed to start the exercise program immediately, while the rest became the wait-list control.
Masking Description: Masking is not practical for an exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise (Experimental): Pilates exercise, Trying to do 25 min of Pilates 3x/week for 8 wks
  Interventions: Other: Online Pilates exercise
- Wait-list control (No Intervention): Waiting 8 weeks without starting Pilates

INTERVENTIONS:
Other: Online Pilates exercise — Participants will be asked to do their Pilates practice while watching the videos (not from memory) to ensure that they are performing techniques optimally. Each module lasts 25 minutes, but includes some resting activities so modules are not vigorous or fatiguing for most people. Nonetheless, subjects will be instructed to omit activities that they feel they cannot do safely. Participants can pause a session to add more rest breaks, if needed, or stop and complete a session later. Participants will attempt to do 3 Pilates modules per week, for a total of 75-90 minutes/week (depending on the exact length of the modules they do).
  Arms: Pilates exercise

SUMMARY:
People with hypermobile Ehlers-Danlos Syndrome/Hypermobility Spectrum Disorder (hEDS/HSD) often have pain, coordination problems, and low tolerance to activity and exercise. There is a publicly available on-line, independent Pilates program designed specifically for this population. This research project proposes to measure pain, function, and common symptoms in individuals before and after 8 weeks of using this on-line Pilates module, and will follow up 6 months later, and compare to an 8-week wait-list control group.

DETAILED DESCRIPTION:
The intervention is provided through an on-line Pilates module commercially available at https://jeanniedibon.com/strengthen-your-hypermobile-core/. "Strengthen Your Hypermobile Core" has 5 modules. Subjects will be asked to complete the modules in order, as the modules build upon one another. However, subjects may repeat any modules at any time, with the goal of completing all 5 modules within the 8 week period. This allows subjects the flexibility to customize their participation by using the modules they feel are most helpful. Users who typically access this Pilates course have this same flexibility so, while it adds variability to the intervention, it better reflects how the program is actually used.

Subjects will be asked to do their Pilates practice while watching the videos (not from memory) to ensure that they are performing techniques optimally. Each module lasts 25 minutes, but includes some resting activities so modules are not vigorous or fatiguing for most people. Nonetheless, subjects will be instructed to omit activities that they feel they cannot do safely. Subjects can pause a session to add more rest breaks, if needed, or stop and complete a session later. Subjects will commit to doing 3 Pilates modules per week, for a total of 75-90 minutes/week (depending on the exact length of the modules they do).

Subjects will complete questionnaires before starting the on-line Pilates modules. Completing these questionnaires on SurveyMonkey is likely to take 30-45 minutes.

The study initially aimed to include a total of 100 participants, but more than 800 signed up within the first 2 weeks, and another 200 over the following months. The design was therefore modified to have the first 300 participants start the Pilates immediately, and the remaining participants begin after an 8-week waiting period. In addition to adding a control group, the wait-list prevented us from having to turn people away from free access to the exercise program, and from our being overwhelmed by too many participants. Because subjects were not randomly assigned and the intervention could not be directly monitored, the study is a pragmatic clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* i. Have some form of Hypermobility Spectrum Disorders or hypermobile Ehlers-Danlos syndrome (HSD/hEDS) diagnosed by any health care provider; this would include individuals diagnosed with Joint Hypermobility Syndrome using the pre-2017 diagnostic criteria.

ii. Able to read the English language and understand spoken English. iii. Willing to try to do Pilates using the 25 minute on-line training videos at least 3 times per week, unless they experience some adverse event or illness that prevents them from safely participating.

Exclusion Criteria:

* i. Medical restrictions (such as recent and healing surgery, fractures, comorbidities such as severe rheumatoid arthritis or neurological conditions, etc.) that prevent them from safely doing gentle exercise lying down on the floor, sitting, and standing.

ii. Inability to safely stand (with or without using upper extremity for balance) for 10 consecutive minutes.

iii. Recent injuries or changes in status that are not stable. This will be defined as "A significant change in your wellness due to recent injury or new symptoms in the past month that result in your wellness during the past month being very different from the past 5 months. Flare episodes that are typical for you will not prevent you from participating at this time." iv. Significantly changed treatment approach or medication within the past 3 months or be expecting to change their treatment program (including medication changes) during the study. This would make it difficult for us to know if changes are due to the Pilates class or the change in their treatment program. However, we understand that their health status may change such that they need to change their health care routine for physical and mental health.

v. Currently receiving regular rehabilitation such as physical therapy, or having received physical therapy (PT) or a similar movement-based therapy (such as such as Pilates, Feldenkrais, Tai Chi, qigung, yoga) in the past 3 months. Individuals who continue to do exercises from any of these sources are not excluded, as these individuals should be stable on their current routine.

vi. Currently doing more than 30 minutes/week of Pilates exercise.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
Bristol Impact of Hypermobility questionnaire (BIoH) | Enrollment, after 8 weeks of Pilates, 6 months after completed Pilates.
  The BIoH is a 55 item questionnaire that asks about pain, fatigue, joint instability, function, self-efficacy and attitudes about having hypermobility. It is the only outcome measure specifically validated for hypermobility-related conditions, and it is recommended by the international Common Data Elements initiative, whose goal is to encourage Ehlers-Danlos syndrome (EDS) researchers to use consistent outcome measures. (Palmer, 2017)

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK) | Enrollment, after 8 weeks of Pilates, 6 months after completing Pilates.
  Kinesiophobia will be assessed through the Tampa Scale of Kinesiophobia, short form (TSK-11), which is an 11-question survey asking about fear of movement and fear of injury.(Woby, 2005) The Tampa Scale of Kinesiophobia is one of the recommended Common Data Elements for EDS.
The Revised Body Awareness Rating Questionnaire (R-BARQ) | Enrollment, after 8 weeks of Pilates, 6 months after completing Pilates.
  The Revised Body Awareness Rating Questionnaire (R-BARQ) includes 12 questions that ask about body awareness, response to discomfort, breathing patters, and physical response to stress.(Dragesund, 2018) This tool may provide insight into the mechanism by which functional improvements are achieved, by correlating functional improvements with improved body awareness, relaxation, effective breathing, etc.
The International Physical Activity Questionnaire Short Form | Time Frame: Enrollment, after 8 weeks of Pilates, 6 months after completing Pilates.
  The International Physical Activity Questionnaire Short Form is a validated survey assessing physical activity during work, sport, and leisure time. (Booth, 2000)

OTHER OUTCOMES:
Adverse events | After 8 weeks of Pilates
  We asked the question "Have you had any increased pain or problems, beyond mild soreness from doing new exercises, that you think is due to the Pilates?" and the follow-up question "If you have had discomfort related to the Pilates, please briefly describe."

CONTACTS AND LOCATIONS:
Overall Officials: Leslie N. Russek, Principal Investigator — Professor Emeritus
Locations (1):
- Clarkson University. Entire study is online, no physical site used., Potsdam, New York, United States

IPD SHARING:
Plan to Share IPD: No
Hope to share data.

REFERENCES:
- [Background] Booth M. Assessment of physical activity: an international perspective. Res Q Exerc Sport. 2000 Jun;71(2 Suppl):S114-20. No abstract available. PMID 10925833
- [Background] Dragesund T, Strand LI, Grotle M. The Revised Body Awareness Rating Questionnaire: Development Into a Unidimensional Scale Using Rasch Analysis. Phys Ther. 2018 Feb 1;98(2):122-132. doi: 10.1093/ptj/pzx111. PMID 29096009
- [Background] Palmer S, Cramp F, Lewis R, Gould G, Clark EM. Development and initial validation of the Bristol Impact of Hypermobility questionnaire. Physiotherapy. 2017 Jun;103(2):186-192. doi: 10.1016/j.physio.2016.04.002. Epub 2016 May 4. PMID 27567344
- [Background] Woby SR, Roach NK, Urmston M, Watson PJ. Psychometric properties of the TSK-11: a shortened version of the Tampa Scale for Kinesiophobia. Pain. 2005 Sep;117(1-2):137-44. doi: 10.1016/j.pain.2005.05.029. PMID 16055269

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT07118865/Prot_SAP_ICF_000.pdf